CLINICAL TRIAL: NCT05311202
Title: The Effect of Training Volume and Intensity of Acute Resistance Exercise on Inhibitory Control: An Event-Related Potential Study
Brief Title: The Effect of Acute Resistance Exercise on Inhibitory Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yu-Kai Chang, Research Chair professor, National Taiwan Normal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PACNL_202201HM012
Record Dates: First submitted 2022-03-16; First posted 2022-04-05 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Exercise; Cognitive Function
Keywords: Acute resistance exercise; Inhibitory control; Training volume; Intensity; Event-related potential
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- low-volume moderate-intensity group (Experimental): Participants will attend the trainer-supervised resistance exercise program for 30 minutes
  Interventions: Behavioral: low-volume moderate-intensity group
- moderate-volume moderate-intensity group (Experimental): Participants will attend the trainer-supervised resistance exercise program for 40 minutes
  Interventions: Behavioral: moderate-volume moderate-intensity group
- high-volume moderate-intensity group (Experimental): Participants will attend the trainer-supervised resistance exercise program for 50 minutes
  Interventions: Behavioral: high-volume moderate-intensity group
- moderate-volume low-intensity group (Experimental): Participants will attend the trainer-supervised resistance exercise program for 45 minutes
  Interventions: Behavioral: moderate-volume low-intensity group
- Control group (Experimental): Reading for 40 minutes
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: low-volume moderate-intensity group — The interventional program will include (1) 5 minutes of warm-up and aerobic exercise from light to moderate intensity; (2) 20 minutes of two sets of moderate intensity resistance exercise with 10 repetitions; (3) 5 minutes of cool down
  Arms: low-volume moderate-intensity group
Behavioral: moderate-volume moderate-intensity group — The interventional program will include (1) 5 minutes of warm-up and aerobic exercise from light to moderate intensity; (2) 30 minutes of three sets of moderate intensity resistance exercise with 10 repetitions; (3) 5 minutes of cool down
  Arms: moderate-volume moderate-intensity group
Behavioral: high-volume moderate-intensity group — The interventional program will include (1) 5 minutes of warm-up and aerobic exercise from light to moderate intensity; (2) 40 minutes of four sets of moderate intensity resistance exercise with 10 repetitions; (3) 5 minutes of cool down
  Arms: high-volume moderate-intensity group
Behavioral: moderate-volume low-intensity group — The interventional program will include (1) 5 minutes of warm-up and aerobic exercise from light to moderate intensity; (2) 35 minutes of four sets of low intensity resistance exercise with 20 repetitions; (3) 5 minutes of cool down
  Arms: moderate-volume low-intensity group
Behavioral: Control group — Reading a book related to cognitive function & exercise for 40 minutes
  Arms: Control group

SUMMARY:
The current study is a five-arm, single bout program aiming to assess the effects of training volume and intensity of acute resistance exercise on inhibitory control on neurocognitive function with respect to event-related potential in adults aged 20 - 26 years.

DETAILED DESCRIPTION:
The current study is expected that 175 healthy adults will be recruited and randomly assigned to control group, low volume-moderate intensity, moderate volume-moderate intensity, high volume-moderate intensity, or moderate volume-low intensity group, with 35 participants in each group. Participants will be required to conduct two experiments. The first was the familiarity experiment, which consisted of the experiment description, the familiarity test, and the 6 Repetition Maximum (RM) test. The process lasted about 3 hours. The exercise group was given a warm-up exercise before the intervention, followed by resistance exercise, including Bench Press, Rowing, Deadlift, and Squat, all completed on the Smith machine. After the exercise, the group was given a cool down, while the control group was given 30 minutes of reading. Before and after the intervention, Stroop, event-related potential and fingertip blood lactate were measured, and another fingertip blood lactate was measured 10 minutes after the intervention, which lasted about 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* The dominant hand is right-handed
* 18.5 < BMI < 26
* Can cooperate with fingertip blood collection
* No color blindness and epilepsy
* Not taking medications that affect brain function
* Irregular exercise (more than 150 minutes per week for 3 months)

Exclusion Criteria:

* The participants who do not meet the inclusion or The Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) Criteria.

Ages: 20 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes In Inhibitory Control | 30 minutes each before & after intervention
  The computerized Stroop test will be administrated to assess participants' inhibitory function, and the changes in Emotional Stroop test performance (i.e., response time and accuracy) before (pre-test) and after (post-test) intervention will be examined.
Changes In Neuroelectrical Activities: Event-Related Potential Recording and Analysis | 30 minutes each before & after intervention
  The continuous electroencephalogram (EEG) activity of each participant will be recorded throughout the entire Stroop task using a Neuroscan Quick-Cap, with 32 Ag/AgCl electrodes arranged following the international 10-20 system (NeuroScan Inc., El Paso, TX, USA). Changes in the neuroelectrical activities before and after the intervention will be examined. The time windows for each ERP component will be determined based on a visual inspection of the averaged grand waveform.

SECONDARY OUTCOMES:
Changes In Positive & Negative Affect | 5 minutes after pre-test and post-test of Stroop test
  The changes in the Positive & Negative affect after pre-and post-test will be assessed by The Positive and Negative Affect Schedule (PANAS) questionnaire, which is made up of two 10-item scales that assess both positive and negative emotions. Each item is scored on a scale of 1 (not at all) to 5 (very much).
Muscular Fitness Measurements (1RM)-Deadlift | 2 hours on the first day
  The greatest weight an individual is capable of lifting for one repetition (1RM) will be examined using the 6-RM assessment according to the American College of Sports Medicine (ACSM) protocol. There were multiple steps in the resistance exercise assessment process. Warming up at a low intensity for 1 minute will be followed by a 1-minute rest break. For the first set of exercises, each person's workload (lbs) will be increased by 10-20% for lower body exercises. Participants will be told to do 10 repetitions followed by a 2-minute rest break during this step. Following that, a steadily increasing load will be applied until the load can only be completed less than 6 repetitions. The numbers of set will be limited to the minimum 1set to maximum 4sets. The 1RM will be caculated by the results of 6-RM protocol.
Muscular Fitness Measurements (1RM)-Bench Press | 2 hours on the first day
  The greatest weight an individual is capable of lifting for one repetition (1RM) will be examined using the 6-RM assessment according to the American College of Sports Medicine (ACSM) protocol. There were multiple steps in the resistance exercise assessment process. Warming up at a low intensity for 1 minute will be followed by a 1-minute rest break. For the first set of exercises, each person's workload (lbs) will be increased by 5-10%. Participants will be told to do 10 repetitions followed by a 2-minute rest break during this step. Following that, a steadily increasing load will be applied until the load can only be completed less than 6 repetitions. The numbers of set will be limited to the minimum 1set to maximum 4sets. 1RM will be caculated by the results of 6-RM protocol.
Muscular Fitness Measurements (1RM)-Squat | 2 hours on the first day
  The greatest weight an individual is capable of lifting for one repetition (1RM) will be examined using the 6-RM assessment according to the American College of Sports Medicine (ACSM) protocol. There were multiple steps in the resistance exercise assessment process. Warming up at a low intensity for 1 minute will be followed by a 1-minute rest break. For the first set of exercises, each person's workload (lbs) will be increased by 10-20% for. Participants will be told to do 10 repetitions followed by a 2-minute rest break during this step. Following that, a steadily increasing load will be applied until the load can only be completed less than 6 repetitions. The numbers of set will be limited to the minimum 1set to maximum 4sets. 1RM will be caculated by the results of 6-RM protocol.
Muscular Fitness Measurements (1RM)-Rowing | 2 hours on the first day
  The greatest weight an individual is capable of lifting for one repetition (1RM) will be examined using the 6-RM assessment according to the American College of Sports Medicine (ACSM) protocol. There were multiple steps in the resistance exercise assessment process. Warming up at a low intensity for 1 minute will be followed by a 1-minute rest break. For the first set of exercises, each person's workload (lbs) will be increased by 5-10%. Participants will be told to do 10 repetitions followed by a 2-minute rest break during this step. Following that, a steadily increasing load will be applied until the load can only be completed less than 6 repetitions. The numbers of set will be limited to the minimum 1set to maximum 4sets. 1RM will be caculated by the results of 6-RM protocol.
Changes In Concentration Of Blood Lactate | 2 minutes of each time point (Before the pre-test of cognitive test, after the intervention and before the post-test of cognitive test)
  Fingertip Blood samples will be collected using Lactate Analyzer in three times point: before the pre-test of cognitive test, after the intervention and before the post-test of cognitive test, and analysed the change in concentration of blood lactate between the three time points.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, Ph.D., Principal Investigator — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen YC, Lo YH, Hung CS, Cheng YT, Li RH, Chen FT, Chang YK. Acute effects of resistance exercise intensity and repetition at a predetermined volume on inhibitory control: a randomized controlled trial. Front Sports Act Living. 2025 Mar 13;7:1551624. doi: 10.3389/fspor.2025.1551624. eCollection 2025. PMID 40181929